CLINICAL TRIAL: NCT05700695
Title: Intravenous Branched-chain Amino Acids for Overt Hepatic Encephalopathy in Patients With Acute on Chronic Liver Failure - A Multi-centric Double-blind Randomized Controlled Trial
Brief Title: Intravenous BCAA for HE in ACLF (BCAA-HE-ACLF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Amrita Institute of Medical Sciences & Research Center (Other); Asian Institute of Gastroenterology, India (Other); All India Institute of Medical Sciences, Bhubaneswar (Other); Kalinga Institute of Medical Sciences, Bhubaneswar (Unknown)
Responsible Party: Principal Investigator, Madhumita Premkumar, ASSOCIATE PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC/04/2022-2385
Record Dates: First submitted 2022-12-06; First posted 2023-01-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure
Keywords: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Neurological Dysfunction; Metabolomics; Systemic Inflammations; Branch Chain Amino Acid; bispectral index; Cerebral edema; Lactulose
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure; Brain Edema | interventions — Amino Acids; Lactulose

STUDY DESIGN:
Intervention Model Description: Prospective interventional cohort study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Placebo Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experiential Arm (Experimental): Drug: iv Branch Chain Amino Acid + Lactulose Intravenous Branched Chain Amino Acids - 500mL once daily for 3 days plus Lactulose
  Interventions: Drug: Branch Chain Amino Acid; Drug: Lactulose
- Comparator Arm (Active Comparator): Drug: Lactulose + Placebo of IV BCAA solution
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Branch Chain Amino Acid — Intravenous branched chain amino acids will be given for 3 days to patients in experimental arm
  Arms: Experiential Arm
Drug: Lactulose — Oral lactulose will be given to patients in both arms

SUMMARY:
This multi-centric study analyses the effect of intravenous branched-chain amino acids (BCAA) on overt HE in patients with ACLF. The investigators aim to study the efficacy of combining intravenous BCAA with lactulose versus lactulose alone, ammonia measures, endotoxin, metabolomics, and cerebral edema in the medical management of overt HE in patients with ACLF. The study will also access the impact on overall survival and improvement in the grade of HE.

DETAILED DESCRIPTION:
Treatment of HE in ACLF is based on extrapolation of data available from cirrhotic patients with HE. The mainstay of treatment remains Lactulose. Rifaximin is added on to therapy who have a breakthrough episode of HE on lactulose. BCAA is used as an add-on therapy if patients have minimal/covert encephalopathy, are protein intolerant or have recurrent HE. No studies are available assessing the adjuvant effect of intravenous BCAA on ammonia reduction in HE in patients with ACLF. So, this study has been designed to analyze the effect of intravenous BCAA on hepatic encephalopathy in patients with ACLF. This study will also analyze the systemic and neuronal inflammation, metabolomics, and cerebral edema under the effect of intravenous BCAA in HE patients with ACLF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Either gender
3. Patients with ACLF (CANONIC definition) of any etiology with HE ≥grade 2 as per West-Haven Criteria

Exclusion Criteria:

1. Those who do not consent to participate in the study
2. Patients with structural brain lesions or stroke
3. Inability to obtain informed consent from patient or relatives
4. Severe preexisting cardiopulmonary disease
5. Renal dysfunction (S. Creatinine ≥ 2mg/dL)
6. Pregnancy/Lactation
7. Post liver transplant patients
8. HIV infection
9. Patients who are on psychoactive drugs, like sedatives or antidepressants
10. Patients who are too sick to carry out the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Survival | Day 28
  Survival assessment will be made by recording all deaths

SECONDARY OUTCOMES:
Reduction of arterial ammonia Level | Day 3
  Level of ammonia will be measured by Point of care device
Reduction of arterial ammonia Level | Day 7
  Level of ammonia will be measured by Point of care device
Assessment of cerebral edema | Discharge form Hospital and 3 month of episode of HE
  Cerebral edema will be assessed by Magnetic Resonance Imaging+ Magnetic Resonance Spectroscopy
Prevention/reduction of cerebral edema based on optic nerve sheath diameter (ONSD) | 72 Hours
  ONSD measurement will be done by Ultrasound
Reduction of consciousness recovery time among survivors | Day 28
  Consciousness will be assessed by cognitive battery tests
Survival | Day 28
  Survival assessment will be done with recording all cause mortality
Survival | Day 90
  Survival assessment will be done with recording all cause mortality
Improvement of encephalopathy by one or more grade | Day 7
  Improvement in scoring of hepatic Encephalopathy
Assessment of metabolomics following BCAA + Lactulose and Lactulose alone | Day 7
  Metabolomics will be performed by LC/GC-MS
Dynamic Assessment of systemic inflammation (Cytokines: IL-1b, IL-6, INF-g, TNF-a, IL-15, IL-17, IL-18) at presentation and after Specific management. | Day 0
  Systemic inflammation will be accessed by Cytometric Bead Array

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Madhumita Premkumar, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shawcross DL, Sharifi Y, Canavan JB, Yeoman AD, Abeles RD, Taylor NJ, Auzinger G, Bernal W, Wendon JA. Infection and systemic inflammation, not ammonia, are associated with Grade 3/4 hepatic encephalopathy, but not mortality in cirrhosis. J Hepatol. 2011 Apr;54(4):640-9. doi: 10.1016/j.jhep.2010.07.045. Epub 2010 Dec 1. PMID 21163546
- [Background] Norenberg MD, Martinez-Hernandez A. Fine structural localization of glutamine synthetase in astrocytes of rat brain. Brain Res. 1979 Feb 2;161(2):303-10. doi: 10.1016/0006-8993(79)90071-4. PMID 31966
- [Background] Albrecht J, Norenberg MD. Glutamine: a Trojan horse in ammonia neurotoxicity. Hepatology. 2006 Oct;44(4):788-94. doi: 10.1002/hep.21357. PMID 17006913
- [Background] Donovan JP, Schafer DF, Shaw BW Jr, Sorrell MF. Cerebral oedema and increased intracranial pressure in chronic liver disease. Lancet. 1998 Mar 7;351(9104):719-21. doi: 10.1016/S0140-6736(97)07373-X. PMID 9504517
- [Background] Laake JH, Takumi Y, Eidet J, Torgner IA, Roberg B, Kvamme E, Ottersen OP. Postembedding immunogold labelling reveals subcellular localization and pathway-specific enrichment of phosphate activated glutaminase in rat cerebellum. Neuroscience. 1999;88(4):1137-51. doi: 10.1016/s0306-4522(98)00298-x. PMID 10336125
- [Background] Fischer JE, Rosen HM, Ebeid AM, James JH, Keane JM, Soeters PB. The effect of normalization of plasma amino acids on hepatic encephalopathy in man. Surgery. 1976 Jul;80(1):77-91. PMID 818729
- [Background] Rossi-Fanelli F, Riggio O, Cangiano C, Cascino A, De Conciliis D, Merli M, Stortoni M, Giunchi G. Branched-chain amino acids vs lactulose in the treatment of hepatic coma: a controlled study. Dig Dis Sci. 1982 Oct;27(10):929-35. doi: 10.1007/BF01316578. PMID 6749458
- [Background] Cordoba J, Ventura-Cots M, Simon-Talero M, Amoros A, Pavesi M, Vilstrup H, Angeli P, Domenicali M, Gines P, Bernardi M, Arroyo V; CANONIC Study Investigators of EASL-CLIF Consortium. Characteristics, risk factors, and mortality of cirrhotic patients hospitalized for hepatic encephalopathy with and without acute-on-chronic liver failure (ACLF). J Hepatol. 2014 Feb;60(2):275-81. doi: 10.1016/j.jhep.2013.10.004. Epub 2013 Oct 12. PMID 24128414
- [Background] Dam G, Aamann L, Vistrup H, Gluud LL. The role of Branched Chain Amino Acids in the treatment of hepatic Encephalopathy. J Clin Exp Hepatol. 2018 Dec;8(4):448-451. doi: 10.1016/j.jceh.2018.06.004. Epub 2018 Jun 27. PMID 30568347
- [Background] Gluud LL, Dam G, Les I, Cordoba J, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2015 Feb 25;(2):CD001939. doi: 10.1002/14651858.CD001939.pub2. PMID 25715177
- [Background] Bajaj JS, Wade JB, Sanyal AJ. Spectrum of neurocognitive impairment in cirrhosis: Implications for the assessment of hepatic encephalopathy. Hepatology. 2009 Dec;50(6):2014-21. doi: 10.1002/hep.23216. No abstract available. PMID 19787808